CLINICAL TRIAL: NCT05504668
Title: The Cognitive Effects of 'Brainwaves' Supplementation in Cognitively Intact Older Adults Experiencing Subjective Memory Decline: A Randomized, Placebo Controlled, Parallel Groups Investigation
Brief Title: The Cognitive Effects of 'Brainwaves' Supplementation in Cognitively Intact Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Pukka Herbs Limited (Unknown)
Responsible Party: Principal Investigator, Emma Wightman, Associate Professor, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 50BP1
Record Dates: First submitted 2022-08-16; First posted 2022-08-17 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Cognitive Change; Mood Change; Microbial Colonization
Keywords: Turmeric; Cognition; Microbiome; Metabolome
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind with a placebo control. The study funder organised the formulation of both the active and placebo capsules originally in 2019 so that they were aesthetically identical. Approximately half-way through the trial, the treatments expired due to Covid-19-induced delays and the remainder of the products required to complete the trial were reconstituted by staff at Northumbria University who had no further involvement in the trial. Capsules were again matched to be aesthetically identical between active and placebo but these treatments looked different to those in the first portion of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Turmeric Brainwave (Experimental): Turmeric Brainwaves (now Mind Focus) is a proprietorial herbal supplement from Pukka Herbs which contains (inc. mg daily dose when 2 capsules combined); brahmi (320 mg), gotu kola leaf (144 mg), turmeric whole powder (116 mg), reishi full spectrum (116 mg), rosemary (116 mg), cardamom (88 mg), holy basil (86 mg), turmeric Wholistic™ extract (58 mg), green tea (58 mg) and seagreens (58 mg).
  Interventions: Dietary Supplement: Turmeric Brainwave
- Placebo (Placebo Comparator): Magnesium Stearate
  Interventions: Dietary Supplement: Turmeric Brainwave

INTERVENTIONS:
Dietary Supplement: Turmeric Brainwave — A multiingredient herbal supplement with Turmeric as its most abundant single ingredient.

SUMMARY:
This study investigated the effects of a proprietorial herbal supplement, Turmeric Brainwave (now Mind focus), on cognition, mood and the microbiome in older adults experiencing subjective memory decline, following 90 days supplementation.

DETAILED DESCRIPTION:
The primary aim of this randomised, double blind, placebo-controlled, parallel groups study was to assess the effects of a daily dose of Turmeric Brainwaves, versus placebo, both acutely and following 90 days consumption. Effects were to be assessed in 55-75 year old males and females who reported that their memory now was worse than when in their 20's. Effects were assessed via cognitive (including COMPASS and Cognimapp as well as 2 real-world long-term memory tasks (location-action (AKA Prospective Remembering Video Procedure (PRVP)) and recall of facts)) and mood (using visual analogue scales) outcomes and, additionally, stool and urine samples collected at the beginning and the end of the trial period assessed the microfloral community of the gut and urinary metabolome.

ELIGIBILITY:
Inclusion Criteria:

* 55-75 years at time of enrolment
* Answers yes to the question 'would you say that your memory now is worse now than it used to be in your 20's?'

Exclusion Criteria:

* Pre-existing medical condition/illnesses which would impact taking part in the study The explicit exceptions to this were controlled (medicated) arthritis, asthma, hay fever, high cholesterol and reflux-related conditions. Other, unforeseen, exceptions were considered on a case-by-case basis; i.e. participants may have progressed to screening if they had a condition/illness which would not interact with the active treatments or impede performance.
* Currently taking prescription medications The explicit exceptions to this were contraceptive and hormone replacement treatments for female participants where symptoms were stable and treatment would not change during the course of the study, those medications used in the treatment of arthritis, high cholesterol and reflux-related conditions and those taken 'as needed' in the treatment of asthma and hay fever. As above, there may have been other instances of permitted medication use where no interaction with the active treatments was anticipated.
* High blood pressure (BP; systolic over 159 mm Hg or diastolic over 99 mm Hg)
* Body Mass Index (BMI) outside of the range 18.5-30 kg/m2
* Pregnant, seeking to become pregnant or lactating
* Learning and/or behavioural difficulties such as dyslexia or Attention Deficit Hyperactivity Disorder (ADHD)
* Visual impairments not corrected with glasses or contact lenses (including colour-blindness)
* Smoking (including vaping)
* Excessive caffeine intake (>500 mg per day)
* Clinically diagnosed food intolerances/sensitivities
* Antibiotic, prebiotic or probiotic (including drinks; e.g. Yakult or Actimel) use within the past 8 weeks
* Health conditions preventing fulfilment of the study requirements (this included non-diagnosed conditions for which no medication was taken)
* Inability to complete all of the study assessments
* Currently participating in other clinical or nutrition intervention studies, or had in the past 4 weeks (8 weeks if a probiotic study)
* Diagnosed with/ undergoing treatment for alcohol or drug abuse in the last 12 months
* Diagnosed with/ undergoing treatment for a psychiatric disorder in the last 12 months
* Suffering from frequent migraines that require medication (more than or equal to 1 per month)
* Sleep disturbances (including night-shift work) and/or are taking sleep aid medication
* Any known active infections
* Does not have a bank account (required for payment)
* Are non-compliant with regards treatment consumption

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Cognitive function (lab-based) | 90 days
  This outcome will be assessed via changes on the cognitive task outcomes (measured via COMPASS). COMPASS is a proprietorial software platform for delivering a range of cognitive tasks; assessing domains like memory and attention, with tasks scored for accuracy (% correct) and speed (msec).

SECONDARY OUTCOMES:
Cognitive function (remote) | 90 days
  This outcome will be assessed via changes on the cognitive task outcomes (measured via Cognimapp). Cognimapp is a proprietorial software platform for delivering a range of cognitive tasks via mobile phone; assessing domains like memory and attention, with tasks scored for accuracy (% correct) and speed (msec).
Mood (Anxiety) | 90 days
  This outcome will be assessed via changes on the Generalised Anxiety Disorder 7 (GAD 7) questionnaire. This questionnaire comprises 7 items which are scored from 0 (not at all) to 3 (nearly every day) with a higher score indicating greater anxiety.
Mood (General) | 90 days
  This outcome will be assessed via changes on Visual Analogue Scales (VAS). This VAS is a 100 mm line with mood related adjectives anchoring each end of the line. This is scored from mm distance along the line; with a higher score indicating greater feeling of that mood facet.
Prospective memory | 90 days
  This facet of memory is assessed by the Prospective Remembering Video Procedure (PRVP) which is an 18-item list of locations and actions depicted within a 10-minute video. Participants must encode these locations and actions and recall them when watching this video at a later date.
Delayed recall | 90 days
  This is a real-world recall of 10 facts, created by the principal investigator for the purposes of this study, which participants encode at the start of the trial and must recall at the end.
Gut microbiota | 90 days
  This will be assessed by any shifts in gut microbial species from a stool sample collected at the start of the trial compared to the stool sample taken at the end.
Urinary metabolome | 90 days
  This will be assessed by any shifts in markers identified within the urinary metabolome from a urine sample collected at the start of the trial compared to the urine sample taken at the end.

CONTACTS AND LOCATIONS:
Overall Officials: Emma L Wightman, PhD, Principal Investigator — Northumbria University
Locations (1):
- Brain Performance and Nutrition Research Centre, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No
It is likely that we will make the data available upon request, via email, to the principal investigator but this still needs to be confirmed.

REFERENCES:
- [Derived] Wightman E, Khan J, Smith E, Rolfe V, Smith D, Young G, Cheung W, Kennedy D. Chronic supplementation of a multi-ingredient herbal supplement increases speed of cognitive task performance alongside changes in the urinary metabolism of dopamine and the gut microbiome in cognitively intact older adults experiencing subjective memory decline: a randomized, placebo controlled, parallel groups investigation. Front Nutr. 2023 Oct 10;10:1257516. doi: 10.3389/fnut.2023.1257516. eCollection 2023. PMID 37885445